CLINICAL TRIAL: NCT03937544
Title: A Phase II/III Prospective, Open Label Study to Evaluate Safety and Efficacy of Intravenous Autologous CD19 CAR-T Cells for Relapsed/ Refractory B-Acute Lymphoblastic Leukaemia
Brief Title: Intravenous Autologous CD19 CAR-T Cells for R/R B-ALL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Gaia Science (Other)
Responsible Party: Principal Investigator, Prof. Dr S Fadilah Abdul Wahid, Head of Pusat Terapi Sel / Principal Investigator, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2019-003; FF-2019-138 (Other: UKM Medical Centre)
Record Dates: First submitted 2019-04-22; First posted 2019-05-03 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Relapsed B Acute Lymphoblastic Leukaemia; Refractory B Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T CELLS (Experimental): A conditioning chemotherapy regiment of fludarabine and cyclophosphamide will be administered followed by a single infusion of CAR transduced autologous T cells administered intravenously.
  Interventions: Biological: CD19 CAR-T CELLS; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CD19 CAR-T CELLS — CD19 CAR-T cells will be administered after completion of the lymphodepletion chemotherapy.
Drug: Cyclophosphamide — Patients will receive lymphodepleting chemotherapy consisting of Cyclophosphamide 250 - 300 mg/m2/day IV(Day -5, Day -4, Day -3 ).
Drug: Fludarabine — Patients will receive lymphodepleting chemotherapy consisting of Fludarabine 25-30 mg/m2/day IV (Day -5, Day -4, Day -3 ).

SUMMARY:
This is Phase II / III, Prospective, single arm, Open Label Study to Evaluate Safety and Efficacy of Intravenous Autologous CD19 CAR-T Cells for Relapsed / Refractory B-Acute Lymphoblastic Leukaemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory B-ALL in accordance with World Health Organization (WHO) classification by virtue of BM morphology, flow cytometry, cytogenetics and molecular genetics
* Age between ≥13 to ≤ 65 years
* No detectable leukaemia in the CSF (CNS-1)
* CNS leukaemia without clinically evident neurological symptoms (CNS-2; with <5 WBC per μL and cytology positive for blasts)
* Adequate organ function as defined by a creatinine clearance > 50 ml/min, serum total bilirubin < 5 times the normal value, left ventricular ejection fraction > 40%
* ECOG performance status ≤ 2
* Life expectancy > 3 months
* Post allogeneic HSCT must be ≥ Day +100 with no evidence of active GVHD and not receiving immunosuppression
* Female patients of child bearing age must have negative pregnancy test and is on highly effective contraception methods
* Male patients must use highly effective contraception methods

Exclusion Criteria:

* Patients with CNS-3 leukaemia.
* Active cancer (other than B-ALL).
* Evidence of severe lung, heart (NYHA class III/IV, arrhythmia, AV block, uncontrolled hypertension), liver, or renal failure or severe neurologic disorder.
* Presence of active autoimmune disease or atopic allergy.
* HIV serology positivity.
* Active Hepatitis B or C infection as evidenced by quantitative viral PCR assay.
* Uncontrolled sepsis
* Pregnant / nursing female.
* Ongoing prednisolone > 1mg/kg daily or equivalent.
* Chemotherapy immunotherapy in the recent 4 weeks such as allogeneic cellular therapy weeks, anti-GVHD therapy.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Participants will be followed for the duration of the treatment, with an expected average of 3 months.
  Overall Response Rate (ORR) defined as Complete Response (CR) and CR with incomplete blood recovery (CRi) according to WHO criteria.
Complete response (CR) | 12 Months
  Duration of response defined from the time when criteria for response (CR or CRi) are met to the first documentation of relapse or progression.
CR with incomplete blood recovery (CRi). | 12 Months
  Duration of response defined from the time when criteria for response (CR or CRi) are met to the first documentation of relapse or progression.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 Months, 24 Months
  Overall Survival (OS) defined as the time from treatment to the date of death due to any cause.
Progression free survival (PFS) | 12 Months, 24 Months
  Progression Free Survival (PFS) defined as the time from treatment to first documentation of objective leukemic progression (date of leukaemia assessment documenting progressive disease) or to death due to any cause. Progression is assessed by BM biopsy or CSF analysis according to NCCN criteria. It is assessed at Day 30 and monthly thereafter, or earlier if clinically indicated.
Time to next treatment (TTNT) | 12 Months, 24 Months
  Time To Next Treatment (TTNT) defined as the end of study treatment until the institution of the next therapy.
Percentage of adverse events | 30 days
  Percentage of participants with adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- UKM Medical Centre, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided